CLINICAL TRIAL: NCT02577107
Title: An Exploratory Single Site, Open Label, Randomized, Controlled Study to Evaluate Plasma Vascular Endothelial Growth Factor Levels After Intravitreal Injection of Ranibizumab (Lucentis) and Conbercept (Langmu) for nAMD
Brief Title: Head to Head Study of Anti-VEGF Treatment.
Acronym: RELIANCE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CRFB002ACN07
Record Dates: First submitted 2015-07-30; First posted 2015-10-16 (Estimated); Results first posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-07

CONDITIONS: Age-related Macular Degeneration
Keywords: Age-related macular degeneration,; ranibizumab,; conbercept,; plasma VEGF; PK
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab; KH902 fusion protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ranibizumab 0.5 mg (Experimental): Three monthly injections of 0.5mg Ranibizumab
  Interventions: Drug: ranibizumab
- Conbercept 0.5 mg (Active Comparator): Three monthly injections of 0.5mg Conbercept
  Interventions: Drug: Conbercept

INTERVENTIONS:
Drug: ranibizumab
  Other Names: Lucentis
  Arms: Ranibizumab 0.5 mg
Drug: Conbercept
  Other Names: Langmu
  Arms: Conbercept 0.5 mg

SUMMARY:
An exploratory single site, open label, randomized, controlled study evaluated plasma vascular endothelial growth factor levels after intravitreal injection of ranibizumab (Lucentis) and conbercept (Langmu) for neovascular age-related macular degeneration

DETAILED DESCRIPTION:
This prospective, randomized, open label study enrolled patients with neovascular AMD who were naïve to anti-VEGF therapy or have not received intravitreal anti-VEGF therapy for the previous 3 months. Patients were randomized in two treatment arms for 3 months:

* Study arm 1: Three monthly injections of 0.5mg Ranibizumab
* Study arm 2: Three monthly injections of 0.5mg Conbercept Blood sample (plasma/serum) was collected at baseline (pre-dose), 3h post-injections and days 1, 3, 7 and 28, following doses 1 and 3 for PK and systemic VEGF analysis. The lab staff was blinded for treatment allocation.

Plasma VEGF concentration was measured by a blinded laboratory using Quantikine® ELISA kits. Serum ranibizumab and conbercept concentration will be determined using validated ELISA assay.

The study was divided into 2 stages: the 1st initial feasibility stage with 6 patients per arm (12 patients in total) to verify SD for sample size justification and 2nd stage to confirm the findings with justified sample size.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Male or female patient ≥ 50 years of age.
3. Subfoveal CNV secondary to nAMD.
4. BCVA score must be between 73 and 24 letters as measured by ETDRS chart

Exclusion Criteria:

For both eyes

1. Any active periocular or ocular infection or inflammation
2. Uncontrolled glaucoma
3. Neovascularization of the iris or neovascular glaucoma. For study eye
4. Choroidal neovascularization of any other cause than wet AMD
5. Ocular disorders present that may confound interpretation of study results,
6. Previous treatment with verteporfin PDT (Visudyne®), external-beam radiation therapy, focal laser photocoagulation, vitrectomy, submacular surgery, or transpupillary thermotherapy.
7. Structural damage within 0.5 disc diameter of the center of the macula
8. Atrophy or fibrosis involving the center of the fovea.
9. Inability of obtaining required lab report. Ocular medical history
10. History of intravitreal injection with any anti-VEGF drugs within 3 months. Exclusion criteria for systemic medical conditions and treatment
11. Any type of systemic disease or its treatment
12. Any patients diagnosed with tumor.
13. Stroke or myocardial infarction less than 3 months.
14. Known hypersensitivity to indocyanine green, fluorescein, or any component of the investigational drug formulation.
15. Use of any systemic anti-VEGF drugs within 6 months. Exclusion criteria for patient
16. Patients who have participated in other investigational drug study within 60 days.
17. Pregnant or nursing (lactating) women.
18. Inability to comply with study or follow-up procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2016-07-09 (Actual); Study Completion 2016-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ranibizumab 0.5 mg | Conbercept 0.5 mg
Started | 6 | 6
Completed | 6 | 5
Not Completed | 0 | 1
Not completed — Protocol deviation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab 0.5 mg | Conbercept 0.5 mg | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (5.50) | 69.3 (8.41) | 67.3 (7.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Plasma Vascular Endothelial Growth Factor (VEGF) Concentration After First Injection at Visit 5 (Day 8 +/- 1 Day)
Description: Change from baseline in plasma Vascular endothelial growth factor (VEGF) concentration after first injection at Visit 5 (Day 8 +/- 1 day).Blood sample was collected for systemic VEGF. VEGF was measured by a blinded laboratory using ELISA kits.
Time Frame: Baseline, Visit 5 (Day 8 +/- 1 day)
Population: Per-protocol Set refers to all subjects who completed the study without any major deviation from the study protocol.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ranibizumab 0.5 mg | Conbercept 0.5 mg
Number analyzed (Participants) | 6 | 5
pg/mL | 5.720 (9.5547) | -25.833 (22.8145)
Statistical Analysis 1: Comparison: Ranibizumab 0.5 mg vs Conbercept 0.5 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 20.314, 95% CI 2-sided [9.618 to 31.011], Standard Error of Mean 4.1613

2. Secondary Outcome: Change From Baseline in Plasma Vascular Endothelial Growth Factor (VEGF) Concentration After Third Injection at Visit 10 (Day 67 +/- 1 Day)
Description: Change from baseline in plasma Vascular endothelial growth factor (VEGF) concentration after third injection at Visit 10 (Day 67 +/- 1 day). Blood sample was collected for systemic VEGF. VEGF will be measured by a blinded laboratory using ELISA kits.
Time Frame: Baseline, Visit 10 (Day 67 +/- 1 day)
Population: Per-protocol Set refers to all subjects who completed the study without any major deviation from the study protocol.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ranibizumab 0.5 mg | Conbercept 0.5 mg
Number analyzed (Participants) | 6 | 5
pg/mL | -0.100 (17.4799) | -22.220 (12.9239)

3. Secondary Outcome: Plasma VEGF Concentration at Baseline, Visit 2, 3, 4, 5, 6 After 1st Injection
Description: Blood sample will be collected for systemic VEGF. VEGF will be measured by a blinded laboratory using ELISA kits. Baseline, Visit Visit 2, 3, 4, 5, 6 after 1st injection
Time Frame: Baseline, Visit 2, 3, 4, 5, 6
Population: Per-protocol Set refers to all subjects who completed the study without any major deviation from the study protocol.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ranibizumab 0.5 mg | Conbercept 0.5 mg
Number analyzed (Participants) | 6 | 5
pg/mL
  Baseline | 31.400 (6.3816) | 42.200 (23.4269)
  Visit 2 (Day 1) | 30.958 (19.9813) | 14.920 (12.4920)
  Visit 3 (Day 2 +/- 1) | 36.517 (19.2783) | 24.590 (39.2435)
  Visit 4 (Day 4 +/- 1) | 29.150 (5.5587) | 7.213 (4.9250)
  Visit 5 (Day 8 +/- 1) | 37.000 (4.7979) | 19.075 (4.5051)
  Visit 6 (Day 30 +/- 4) | 27.092 (13.2356) | 25.270 (15.0967)

4. Secondary Outcome: Plasma VEGF Concentration at Baseline, Visit 7, 8, 9, 10, 11 After 3rd Injection
Description: Blood sample will be collected for systemic VEGF. VEGF will be measured by a blinded laboratory using ELISA kits. Baseline, Visit 7, 8, 9, 10, 11 after 3rd injection
Time Frame: Baseline, Visit 7, 8, 9, 10, 11
Population: Per-protocol Set refers to all subjects who completed the study without any major deviation from the study protocol.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ranibizumab 0.5 mg | Conbercept 0.5 mg
Number analyzed (Participants) | 6 | 5
pg/mL
  Baseline | 36.250 (11.8610) | 36.520 (19.2278)
  Visit 7 (Day 60 +/- 4) | 34.383 (12.7727) | 5.720 (2.1690)
  Visit 8 (Day 61 +/- 1) | 46.533 (48.1293) | 6.820 (4.6287)
  Visit 9 (Day 63 +/- 1) | 54.067 (40.2585) | 8.070 (4.6452)
  Visit 10 (Day 67 +/- 1) | 36.150 (25.4399) | 14.300 (9.6690)
  Visit 11 (Day 90 +/- 4) | 45.067 (18.0828) | 56.020 (27.0819)

ADVERSE EVENTS:
Time Frame: Adverse events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All adverse events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit.
Arm/Group | Ranibizumab 0.5 mg | Conbercept 0.5 mg
Serious Adverse Events (participants affected / at risk) | 0/6 | 2/6
Other Adverse Events (participants affected / at risk) | 1/6 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg (N=6) | Conbercept 0.5 mg (N=6)
Infectious pneumonia (Infections and infestations) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Fracture of jaw (Injury, poisoning and procedural complications) | 0 | 1
Fracture of rib (Injury, poisoning and procedural complications) | 0 | 1
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 1
Thoracic injury (Injury, poisoning and procedural complications) | 0 | 1
COPD (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg (N=6) | Conbercept 0.5 mg (N=6)
Dizziness (Ear and labyrinth disorders) | 0 | 1
Conjunctival congestion (Eye disorders) | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 1
Headache (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.